CLINICAL TRIAL: NCT07074847
Title: Coronary Arterial Microcirculation and Metabolism
Status: Enrolling by invitation | Type: Observational
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SPPH-311-320
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Coronary Atherosclerosis of Native Coronary Artery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Measure QFR — Collect blood samples from 100 patients with normal coronary angiography or stenosis less than 50%, centrifuge and collect plasma, and then send them for further metabolomics testing to analyze the test results.

SUMMARY:
Coronary microcirculation disorder refers to a disease in which small blood vessels in the coronary arteries are damaged or blocked, leading to myocardial ischemia and hypoxia. This disease usually occurs in patients with coronary heart disease, but it can also occur in other populations. It is caused by abnormal endothelial function of coronary arteries or spasm of small arteries. Its symptoms include chest pain, shortness of breath, palpitations, etc., which usually occur during physical activity or emotional excitement. If left untreated, it may lead to serious consequences such as myocardial infarction.

The methods for treating coronary microcirculation disorders include drug therapy, surgical treatment, and lifestyle changes. Drug therapy includes antiplatelet drugs, lipid-lowering drugs, vasodilators, etc; Surgical treatment includes coronary artery bypass grafting and percutaneous coronary intervention. Lifestyle changes include quitting smoking, weight control, and increasing physical activity. In summary, coronary microcirculation disorders are a disease that leads to myocardial ischemia and require sufficient attention. Early detection and effective treatment measures can prevent the occurrence of complications and improve the quality of life.

If patients with coronary microcirculation disorders can be detected early and treated accordingly, serious consequences can be avoided. Therefore, we plan to investigate the correlation between coronary microcirculation and metabolomics, with the aim of identifying metabolites closely related to coronary microcirculation from the perspective of metabolomics, in order to elucidate the metabolic processes involved in coronary microcirculation disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal coronary angiography or stenosis less than 50%

Exclusion Criteria:

* Coronary angiography indicates patients with coronary stenosis greater than 50%.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with normal coronary angiography or stenosis less than 50%
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Microcirculatory resistance index | 2025.2.28-2025.12.31

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Shaanxi Provincial People's Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes